CLINICAL TRIAL: NCT03037593
Title: A Randomized Single-Center Study of the Effects of High-Dose Cholecalciferol to Reduce the Incidence of Gestational Diabetes in High-Risk Pregnant Women
Brief Title: High Dose Cholecalciferol to Reduce the Incidence of Gestational Diabetes in High Risk Pregnant Women
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Failure to recruit adequate patients
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1611M98781
Record Dates: First submitted 2017-01-27; First posted 2017-01-31 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Gestational Diabetes
Keywords: Pregnancy; Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: This will be a randomized single-center study with a target study group of 300 women. Women will be followed from enrollment through the remainder of their pregnancy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 4000 IU vitamin D3 +prenatal vitamin
  Interventions: Drug: 4000 IU vitamin D3
- Control (No Intervention): standard prenatal vitamin

INTERVENTIONS:
Drug: 4000 IU vitamin D3 — vitamin D supplementation (4000 IU vitamin D3 +prenatal vitamin
  Other Names: cholecalciferol
  Arms: Intervention

SUMMARY:
Demonstrate dose-dependent relationship between vitamin D supplementation and rates of gestational diabetes.

DETAILED DESCRIPTION:
Determine the effect of increased vitamin D supplementation (4000 IU vitamin D3 +prenatal vitamin) on the incidence of gestational diabetes compared to a standard prenatal vitamin among pregnant women at high risk for gestational diabetes.

Explore the effect of increased vitamin D supplementation (4000 IU daily + prenatal vitamin), compared to a standard prenatal vitamin, on glycemic control, need for oral hypoglycemic agents and/or insulin, and delivery outcomes among the subset of women who develop gestational diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Women who are currently pregnant and receiving prenatal care at the Women's Health Specialists Clinic (University of Minnesota Physicians) from either MD/DO or CNM providers
2. Subject established prenatal care no later than the completed 12th week of gestation (12 6/7 weeks)
3. Subject possesses as least one of the following characteristics:

   1. BMI greater than or equal to 30 kg/m2
   2. History of gestational diabetes in a prior pregnancy
   3. History of infant with birth weight of 4500g or greater
4. Subject is capable of giving informed consent

Exclusion Criteria:

1. Age less than 18 years
2. Multiple gestation pregnancies (twins, triplets or greater multiples)
3. Vitamin D deficiency (defined as less than 20 ng/mL)
4. Preexisting diabetes mellitus defined as either:

   1. pre-existing diagnosis prior to current pregnancy
   2. failure of three-hour glucose tolerance test in first trimester of pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
incidence of gestational diabetes | Baseline to Delivery of child
  effect of increased vitamin D supplementation (4000 IU vitamin D3 +prenatal vitamin) on the incidence of gestational diabetes compared to a standard prenatal vitamin among pregnant women at high risk for gestational diabetes.

SECONDARY OUTCOMES:
Prescription for insulin or oral hypoglycemic agents | Baseline to Delivery of child
  Prescription for insulin or oral hypoglycemic agents
Mode of delivery | Delivery of child
  Natural or C-Section
Birth weight | Delivery of Child
  Weight in Kg
Apgar score | Birth of child to 5 minutes
  <7 at 5 minutes
Shoulder Dystocia | Birth of child

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Hoffman, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Medical Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided